CLINICAL TRIAL: NCT04310904
Title: Cardiac Output Assessment by Using Saline Contrast Injection
Acronym: CardioLog
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0057
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Echocardiography
Keywords: echocardiography; Doppler cardiac output; contrast; thermodilution; agitated saline; ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU cardiac output (CO) assessment patients: all ICU patients intubated/ventilated with a central line and an arterial catheter who need trans esophageal echocardiography examination with a saline contrast test.
  Interventions: Other: contrast assessment of cardiac output (CO); Other: cardiac Doppler technique

INTERVENTIONS:
Other: contrast assessment of cardiac output (CO) — Patients hospitalized in ICU will be included if they need a trans esophageal echocardiographic evaluation and a research of intra cardiac shunt (using a saline contrast test). Patients with Swan Ganz catheter will be included as well. Cardiac output will be measured using cardiac Doppler. Simultaneously, 4.5 ml of saline with 0.5 ml of air will be agitated to have a contrast solution. This solution will be injected as usual and echocardiographic imaging will be recorded. These imaging will be analyzed off-line and CO will be calculated with an algorithm previously developed and compared with the reference method. In case of swan ganz catheter, the cardiac output will be also measured using the thermodilution technique.
Other: cardiac Doppler technique — Patients hospitalized in ICU will be included if they need a trans esophageal echocardiographic evaluation and a research of intra cardiac shunt (using a saline contrast test). Patients with Swan Ganz catheter will be included as well. Cardiac output will be measured using cardiac Doppler. Simultaneously, 4.5 ml of saline with 0.5 ml of air will be agitated to have a contrast solution. This solution will be injected as usual and echocardiographic imaging will be recorded. These imaging will be analyzed off-line and CO will be calculated with an algorithm previously developed and compared with the reference method. In case of swan ganz catheter, the cardiac output will be also measured using the thermodilution technique.

SUMMARY:
Cardiac output (CO) assessment is one of the cornerstone of hemodynamic evaluation in ICU patients. CO is usually measured using invasive methods or non-invasive methods. Thermodilution is considered as the gold standard for CO assessment. Cardiac Doppler as well demonstrated to be accurate but needs manipulations and good knowledge and skills. The investigators developed a new technique using injection of agitated saline solution to evaluate CO without any manual measurement and then observer independent.

DETAILED DESCRIPTION:
The investigators decided to conduct a prospective observational study to compare contrast assessment of CO and cardiac Doppler technique. Patients hospitalized in ICU will be included if they need a trans esophageal echocardiographic evaluation and a research of intra cardiac shunt (using a saline contrast test). Patients with Swan Ganz catheter will be included as well. Cardiac output will be measured using cardiac Doppler. Simultaneously, 4.5 ml of saline with 0.5 ml of air will be agitated to have a contrast solution. This solution will be injected as usual and echocardiographic imaging will be recorded. These imaging will be analyzed off-line and CO will be calculated with an algorithm previously developed and compared with the reference method. In case of swan ganz catheter, the cardiac output will be also measured using the thermodilution technique.

ELIGIBILITY:
Inclusion Criteria:

* all ICU patients intubated/ventilated with a central line and an arterial catheter who need trans esophageal echocardiography examination with a saline contrast test.

Exclusion Criteria:

* patients under 18 years old
* pregnant patients
* moribund patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all ICU patients intubated/ventilated with a central line and an arterial catheter who need trans esophageal echocardiography examination with a saline contrast test.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
variation of cardiac output assessment (CO) | day 0
  correlation will be done between contrast and the reference method cardiac Doppler method.

SECONDARY OUTCOMES:
variation of cardiac output assessment (CO) in patients with a swan gaz catheter | day 0
  comparison will be performed between the contrast CO and the thermodilution CO in the group of patients with a swan ganz catheter

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No